CLINICAL TRIAL: NCT02123498
Title: The Study of the Diagnosis of Eustachian Tube Dysfunction (ETD): Identifying the Relationship of Ear Fullness to Laryngopharyngeal Reflux (LPR)
Brief Title: The Study of Eustachian Tube Dysfunction and Laryngopharyngeal Reflux
Acronym: ETDLPR
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: IRB not approved
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETDLPR2014
Record Dates: First submitted 2014-04-23; First posted 2014-04-25 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2014-04

CONDITIONS: Eustachian Tube Dysfunction; Laryngopharyngeal Reflux
Keywords: ear pressure; ear fullness; ear pain; ETD; laryngopharyngeal reflux; LPR; gastroesophageal reflux disease; GERD; nasopharyngeal reflux; acid reflux
MeSH Terms: conditions — Laryngopharyngeal Reflux; Earache; Gastroesophageal Reflux | interventions — Omeprazole; Ranitidine; Pantoprazole; Laryngoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Omeprazole; Drug: Ranitidine; Drug: Pantoprazole; Procedure: 24-Hour Diagnostic pH-Probe Test; Procedure: Laryngoscopy

INTERVENTIONS:
Drug: Omeprazole — 40mg, to be taken once daily by mouth, 30-60 minutes before meals, for at least 6 weeks
  Other Names: Prilosec
Drug: Ranitidine — 300mg, to be taken once daily by mouth, before bedtime, for at least 6 weeks
  Other Names: Zantac
Drug: Pantoprazole — 40mg, to be taken twice daily by mouth, 30-60 minutes before meals, for at least 6 weeks. (Alternative intervention if participant cannot tolerate omeprazole, is on an anticoagulant medication, or if on medication contraindicated for omeprazole and ranitidine)
  Other Names: Protonix
Procedure: 24-Hour Diagnostic pH-Probe Test — Participants will undergo a routine clinical 24-hour diagnostic pH-probe test to assess quantitative measures for laryngopharyngeal reflux.
Procedure: Laryngoscopy — Participants will undergo routine clinical laryngoscopy to assess presence of laryngopharyngeal reflux.

SUMMARY:
The purpose of this study is to investigate the relationship between ear fullness, pressure, and/or pain and laryngopharyngeal reflux, in order to focus medical therapy and improve therapeutic outcomes in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* They complain of symptoms of ear fullness, ear pain, and/or ear pressure, either unilateral or bilateral
* They are willing to participate in the study.
* They are between the ages of 18 to 80

Exclusion Criteria:

* They have had major ear surgery (not including tympanostomy tubes)
* They have a medical condition that is another possible etiology of ear pain or acid reflux and may require additional medical or surgical intervention such as: Acute or chronic otitis externa, Chronic otitis media, Temporomandibular joint dysfunction, Upper aerodigestive track neoplasm, History of head/neck radiation therapy.
* They are pregnant. Proton pump inhibitors are a Category C drug with unknown pregnancy risks.
* They do not wish to participate in the study
* They are <18 or >80.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Evidence of laryngopharyngeal reflux in patients complaining of ear fullness/pressure/pain | 1 year
  Participants complaining of ear pain, ear fullness, or ear pain are diagnosed with laryngopharyngeal reflux via laryngoscope exam and measurement by diagnostic pH-probe test.

CONTACTS AND LOCATIONS:
Overall Officials: Helen X Xu, MD, Principal Investigator — Loma Linda University Otolaryngology Department
Locations (2):
- United States (2):
  - 11234 Anderson Street, Loma Linda, California
  - 1895 Orange Tree Lane, Suite 102, Redlands, California

REFERENCES:
- [Background] Barbero GJ. Gastroesophageal reflux and upper airway disease. Otolaryngol Clin North Am. 1996 Feb;29(1):27-38. PMID 8834270
- [Background] Crapko M, Kerschner JE, Syring M, Johnston N. Role of extra-esophageal reflux in chronic otitis media with effusion. Laryngoscope. 2007 Aug;117(8):1419-23. doi: 10.1097/MLG.0b013e318064f177. PMID 17585281
- [Background] Heavner SB, Hardy SM, White DR, Prazma J, Pillsbury HC 3rd. Transient inflammation and dysfunction of the eustachian tube secondary to multiple exposures of simulated gastroesophageal refluxant. Ann Otol Rhinol Laryngol. 2001 Oct;110(10):928-34. doi: 10.1177/000348940111001007. PMID 11642425
- [Background] Mims JW. The impact of extra-esophageal reflux upon diseases of the upper respiratory tract. Curr Opin Otolaryngol Head Neck Surg. 2008 Jun;16(3):242-6. doi: 10.1097/MOO.0b013e3282fdc3d6. PMID 18475079
- [Background] Norman G, Llewellyn A, Harden M, Coatesworth A, Kimberling D, Schilder A, McDaid C. Systematic review of the limited evidence base for treatments of Eustachian tube dysfunction: a health technology assessment. Clin Otolaryngol. 2014 Feb;39(1):6-21. doi: 10.1111/coa.12220. PMID 24438176
- [Background] Schreiber S, Garten D, Sudhoff H. Pathophysiological mechanisms of extraesophageal reflux in otolaryngeal disorders. Eur Arch Otorhinolaryngol. 2009 Jan;266(1):17-24. doi: 10.1007/s00405-008-0770-1. Epub 2008 Aug 13. PMID 18704479
- [Background] Yazici ZM, Sari M, Uneri C, Midi A, Tugtepe H. Histologic changes in eustachian tube mucosa of rats after exposure to gastric reflux. Laryngoscope. 2008 May;118(5):849-53. doi: 10.1097/MLG.0b013e318164d0c0. PMID 18300701